CLINICAL TRIAL: NCT04763642
Title: The Comparison of Miniinvasive and Open Pancreaticoduodenectomy for Cancer Pancreaticobiliary Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Budget Public Health Institution Scientific Research Institute - Ochapovsky Regional Clinical Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210202ORCH
Record Dates: First submitted 2021-02-13; First posted 2021-02-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Bile Duct Cancer; Ampulla of Vater Cancer
Keywords: pancreatoduodenectomy; miniinvasive; complication; Morbidity; Mortality
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Laparoscopic Pancreaticoduodenectomy (LPD) (Active Comparator)
  Interventions: Procedure: pancreaticoduodenectomy
- Robotic Pancreaticoduodenectomy (RPD) (Active Comparator)
  Interventions: Procedure: pancreaticoduodenectomy
- Open Pancreaticoduodenectomy (OPD) (Placebo Comparator)
  Interventions: Procedure: pancreaticoduodenectomy

INTERVENTIONS:
Procedure: pancreaticoduodenectomy — Robotic Whipple operation Open Whipple operation Laparoscopic Whipple operation

SUMMARY:
The Comparison of Miniinvasive and Open Pancreaticoduodenectomy for Cancer Pancreaticobiliary Zone

DETAILED DESCRIPTION:
Minimally invasive surgery is undoubtedly the method of choice for multiple gastrointestinal surgical procedures because of its minimally invasive nature and number of benefits such as reducing postoperative pain, shorter hospital stays, and earlier return to work. Current advances in technological innovation and surgical strategies have made surgical procedures on the pancreas a routine practice. However, the use of new surgical techniques in pancreatic surgery has been slow due to the complexity of the operations and the steep learning curve required for their use. For example, minimally invasive pancreatoduodenectomies (MIPD) have not yet become widespread. Due to these interventions have a complex reconstructive stage MIPD are still performed in a very few centers by specialized surgeons.

Although laparoscopic PD was first described in 1994 and the robotic approach in 2003, MIPD still account for less than 14% of all DPE cases. The multicenter randomized controlled trial (LEOPARD-2) for the first time compared laparoscopic and open pancreatoduodenectomy for pancreatic or periampullary tumors. The study that involved 99 patients did not reveal the superiority of laparoscopic PD (LPD) and provided an estimated mortality of 6%; 5 patients died in the laparoscopy group and 1 patient died in the group open PD. The trial was stopped early due to high mortality in the migratory invasive interventions group. Therefore, advantages of minimally invasive procedures for removal of pancreato-biliary zone tumors remain controversial.

In our study, we analyzed perioperative surgical outcomes and short-term survival outcomes in patients undergoing MIPD, including LPD and robotic PD (RPD), as well as "open" proximal pancreatoduodenectomy (OPD).

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-75 years
* Clinically/histologically established diagnosis of the cancer;
* Preoperative imaging assessment is resectable or borderline resectable

Exclusion Criteria:

* Benign tumors of the head of pancreas;
* Distant metastasis;
* Conversion to laparotomy;
* Instrumental findings of the tumor process prevalence;
* General somatic status on the ASA III-V scale;
* Acute pancreatitis;
* Hyperbilirubinemia above 60 μmol/L (3.51 mg/dl) ((normal range, 4-20 μmol/L)).
* Patients with intraoperative positive express-histological presence of tumor growth along the border of the pancreas resection

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Overall complications | up to 30 days
  The proportion of all complications after operation accounted for the total number of patients
Pancreatic fistula | up to 30 days
  The international study group (ISGPF) definition: A drain output of any measurable volume of fluid on or after postoperative day 3 with an amylase content greater than 3 times the serum amylase activity. Three different grades of postoperative fistula (grades A, B, C) are defined according to the clinical impact on the patient's hospital course.
Intra-abdominal bleeding | up to 30 days
  he International Study Group of Pancreatic Surgery (ISGPS) definition: Blood loss through abdominal drains or nasogastric tube;hematemesis or melena; clinical deterioration of the patient; unexplained hypotension or tachycardia; or laboratory findings such as a decreasing hemoglobin concentration.
Intra-abdominal infection | up to 30 days
  Positive cultures of collection of fluid or blood,or persistent fever necessitating treatment with antibiotics and positive detection in image test.

SECONDARY OUTCOMES:
Length of hospital stay (day) | Up to postoperative 2 months
  Participants will be followed for the duration of hospital stay, an expected average of 2 weeks

OTHER OUTCOMES:
progression-free survival | Up to postoperative 3 years
  The period between the beginning of treatment and the observation of disease progression or the occurrence of death for any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Ochapovsky Regional Clinical Hospital № 1, Krasnodar, Krasnodarskiy Kray, Russia

IPD SHARING:
Plan to Share IPD: No